CLINICAL TRIAL: NCT04265807
Title: Remote Ischemic Conditioning to Enhance Resuscitation (RICE) Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Charles F. Kettering Foundation (Unknown)
Responsible Party: Principal Investigator, Graham Nichol, Professor, School of Medicine: Department of Medicine: General Internal Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00005176
Record Dates: First submitted 2020-01-15; First posted 2020-02-12 (Actual); Results first posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Arrest
Keywords: reperfusion injury; remote ischemic conditioning
MeSH Terms: conditions — Heart Arrest; Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Patients and investigators will be masked to treatment assignment up to the point of randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intervention Group (Active Comparator): A standard non-invasive blood pressure cuff (e.g., American Diagnostics Corporation, Hauppauge, NY but any one can be used off the shelf) and disposable plastic clamp (e.g.,Medline Industries Incorporated, Mundelein, IL) can be used to apply RIC in patients resuscitated from OHCA via three cycles of 5-mins. inflation to 200 mmHg followed by 5-mins. deflation of a blood pressure cuff on an upper extremity. The cuff occludes the artery; the clamp maintains pressure in the air bladder of the cuff during the inflation periods.
  Interventions: Device: Active Remote Ischemic Conditioning
- Control Group (Sham Comparator): The control group will have a sham package opened at the bedside as soon as feasible after ED arrival. This will be identical in size, weight and appearance as that in the intervention group, but will contain a sham device. Upon identification that the patient has been randomized to the control group, the care team will proceed with all other resuscitative measures as in the the intervention group.
  Interventions: Device: Sham Remote Ischemic Conditioning

INTERVENTIONS:
Device: Active Remote Ischemic Conditioning — A standard non-invasive blood pressure cuff (e.g., American Diagnostics Corporation, Hauppauge, NY but any one can be used off the shelf) and disposable plastic clamp (e.g.,Medline Industries Incorporated, Mundelein, IL) can be used to apply RIC in patients resuscitated from OHCA via three cycles of 5-mins. inflation to 200 mmHg followed by 5-mins. deflation of a blood pressure cuff on a upper extremity. The cuff occludes the artery; the clamp maintains pressure in the air bladder of the cuff during the inflation periods.
  Arms: Intervention Group
Device: Sham Remote Ischemic Conditioning — The control group will have a sham package opened at the bedside as soon as feasible after ED arrival. This will be identical in size, weight and appearance as that in the intervention group, but will contain a sham device. Upon identification that the patient has been randomized to the control group, the care team will proceed with all other resuscitative measures as in the the intervention group.
  Arms: Control Group

SUMMARY:
Following resuscitation from out-of-hospital cardiac arrest (OHCA), reperfusion injury can cause cell damage in the heart and brain. Remote ischemic conditioning (RIC) consists of intermittent application of a device such as a blood pressure cuff to a limb to induce non-lethal ischemia. Studies in animals with cardiac arrest as well as in humans with acute myocardial infarction suggest that RIC before or after restoration of blood flow may reduce injury to the heart and improve outcomes but this has not been proven in humans who have had OHCA. The RICE pilot study is a single-center study to assess the feasibility of application of RIC in the emergency department setting for patients transported to the hospital after resuscitation from OHCA.

ELIGIBILITY:
Included will be those with:

1. Age 18 years or more;
2. Defibrillation by laypersons or defibrillation and/or chest compressions by EMS providers dispatched to the scene;
3. Non-traumatic etiology of arrest, defined as without concomitant blunt, penetrating, or burn-related injury, or uncontrolled bleeding or exsanguination;
4. Spontaneous circulation upon emergency department arrival;
5. No response to verbal commands; and
6. Ongoing or planned induced hypothermia.

Excluded will be those with:

1. STEMI indicated on first 12-lead ECG obtained after restoration of circulation, defined as ST-elevation of ≥2 mm in two or more contiguous ECG leads;
2. Written do not attempt resuscitation (DNAR) reported to providers before randomization;
3. Drowning or hypothermia as cause of arrest;
4. Known prisoner or pregnant; or
5. Dialysis fistula in either upper extremity; or
6. Pre-existing amputation of upper extremity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graham Nichol, MD, MPH, Principal Investigator — University of Washington; Emilby S Bartlett, MD MS, Principal Investigator — University of Washington
Locations (1):
- Graham Nichol, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Available upon request, subject to mutual agreement
Supporting Information: Study Protocol, CSR

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment occurred from July 01, 2020, to February 03, 2022. Recruitment ceased when target enrollment (30 participants) was achieved. This study was conducted under exception from informed consent (EFIC) for emergency research. Eligible subjects were randomized with masked allocation to control (standard care) versus intervention (standard care and RIC) following OHCA at a single site.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 16 | 14
Completed | 16 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (15.5) | 53.7 (17.4) | 52.5 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 12 | 10 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 10 | 12 | 22
  Unknown or Not Reported | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Attrition
Description: Attrition assessed as the proportion of randomized subjects who do not remain on allocated therapy for the intended study duration among subjects randomly allocated. On therapy for the intended study duration consists of completing three cycles of inflation-deflation.
Time Frame: Completion of their allocated study intervention, an average of 30 minutes from enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 16 | 14
Participants | 0 | 0

2. Secondary Outcome: Treatment Success
Description: Treatment Success assessed as the proportion of intervention group patients who remain alive and on their allocated therapy for the intended study duration.
Time Frame: 30 minutes from initiation of study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 16 | 14
Participants | 16 | 14

3. Secondary Outcome: Cardiac Function
Description: Cardiac Function assessed as left ventricular ejection fraction (LVEF) using echocardiograms ordered for clinical indications.
Time Frame: Within 48 hours of index arrest
Population: This analysis is based on the number of participants with an LVEF recorded.
Measure: Mean (Standard Deviation); unit: % of left ventricular ejection fraction
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 11 | 10
% of left ventricular ejection fraction | 48.4 (20) | 51.7 (12.8)

4. Secondary Outcome: Proportion With Cardiogenic Shock, %
Description: Cardiogenic Shock assessed as systolic BP < 80 mmHg during any 6 h period within 48 h of the index arrest not due to a correctable cause, and treated with pressors or inotropes or placement of a mechanical cardiac assist device (e.g. intra-aortic balloon pump). Cardiogenic shock correlates with survival after resuscitation from cardiac arrest.
Time Frame: Within 48 hours of index arrest
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 16 | 14
Participants | 13 | 11

5. Secondary Outcome: STEMI
Description: STEMI assessed as the presence of electrocardiographic (ECG) and biomarker criteria for acute myocardial infarction within 48 h of the index arrest. Note that ST-elevation on the first 12-lead ECG after resuscitation is a poor predictor of acute infarction in this population. These patients often develop infarctions during the subsequent 48 h.
Time Frame: Within 48 hours of index arrest
Population: One participant in the control group did not have data recorded for this metric (unknown) and was not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 16 | 13
Participants | 0 | 0

6. Secondary Outcome: Myocardial Injury
Description: Myocardial Injury assessed as peak serum troponin in ng/mL at any time point within 24 h of index arrest.
Time Frame: Within 24 hours of index arrest
Population: Participants with an elevated serum troponin (>0.03) were included in the analysis.
Measure: Mean (Standard Deviation); unit: peak serum troponin level
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 15 | 11
peak serum troponin level | 3.7 (8.9) | 7.4 (16.2)

7. Secondary Outcome: Renal Dysfunction
Description: Renal Dysfunction assessed using Risk, Injury, Failure, Loss, End Stage criteria.
Time Frame: Within 24 hours of index arrest
Population: In order to calculate the RIFLE score, both a baseline creatinine level (prior to the index cardiac arrest) and a first recorded creatinine level (after the index cardiac arrest) were required. Only those participants with both creatinine values were included in the analysis. For this analysis, participants with a creatinine level which was 1.5 times above baseline or more were counted as positive for AKI.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 7 | 5
Participants | 4 | 2

8. Secondary Outcome: Hospital Free Survival
Description: Hospital Free Survival (HFS) assessed as number of days alive and permanently out of hospital up to 30 days post arrest
Time Frame: Within 30 days of index arrest
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 16 | 14
days | 11.1 (14.3) | 7.3 (12.3)

9. Secondary Outcome: Withdrawal of Care
Description: assessed as the reduction of support (i.e. reducing pressors, lab draws or medications) or withdrawal of support (i.e. extubation, stopping drips/meds, changing to comfort care only) during hospitalization.
Time Frame: Discharge or 30 days after index arrest
Population: There was missing data on the participants not included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 13 | 13
Participants | 6 | 7

10. Secondary Outcome: Favourable Neurologic Status at Discharge
Description: Favourable Neurologic Status at Discharge assessed using modified Rankin Score (MRS) < 3 at hospital discharge or 30 days after index arrest. Modified Rankin Scale is scored from zero to six. Higher values represent a worse outcome. Favorable neurologic status is defined as a modified Rankin score 0, 1 or 2.
Time Frame: Discharge or 30 days after index arrest
Measure: Median (Inter-Quartile Range); unit: Modified Rankin Score
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 16 | 14
Modified Rankin Score | 6 [1 to 6] | 6 [1.5 to 6]

11. Secondary Outcome: Survival to Discharge
Description: Survival to Discharge assessed as alive when discharged from hospital to home, nursing facility or rehabilitation. Patients transferred to another acute care facility (e.g. to undergo implantable defibrillator placement) will be considered still hospitalized.
Time Frame: Discharge or 30 days after index arrest
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 16 | 14
Participants | 7 | 6

12. Secondary Outcome: Clinical Instability at Discharge
Description: Clinical Instability at Discharge assessed using the Kosecoff Index measured at discharge based on the presence of nine symptoms and signs associated with increased risk of rehospitalization. Instability will be the presence of any of these.
  Clinical instability at discharge was defined by the Kosecoff Index. https://pubmed.ncbi.nlm.nih.gov/2214063/
  This was scored as 1 point for the presence and 0 for the absence of each of the following during the 24 h prior to discharge:
  Fever, temperature >38.3°C Urinary incontinence Chest pain Shortness of breath Confusion Heart rate >=130 beats/min Respiratory rate >=30/min Diastolic blood pressure >= 105 mmHg Systolic blood pressure < 90 mmHg Heart rate < 50 bpm Premature ventricular contractions on telemetry
Time Frame: Discharge or 30 days after index arrest
Population: Participants were included in this analysis if they survived to discharge. Three participants (all from the control group) were missing data on this metric and were also excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 7 | 3
Participants | 3 | 2

13. Secondary Outcome: Survival to 30 Days After Arrest
Description: Survival to 30 Days After Cardiac Arrest assessed as alive 30 days after the index cardiac arrest as confirmed by a brief telephone interview.
Time Frame: 30 days after index arrest
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 16 | 14
Participants | 7 | 6

14. Secondary Outcome: Accrual
Description: Accrual is the proportion of eligible subjects who have the study device applied
Time Frame: Before leaving the emergency department
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 16 | 14
Participants | 16 | 14

15. Other Pre Specified Outcome: Device Failure
Description: device failure will be defined as discontinuation of use of the device prior to the end of allocated treatment interval because of mechanical failure as opposed to provider preference.
Time Frame: 30 minutes from initiation of study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 16 | 14
Participants | 0 | 0

16. Other Pre Specified Outcome: Expected Adverse Event Related to Device- Pain
Description: Pain assessed using the Richmond Agitation-Sedation Scale at 30 and 60 minutes after randomization in control and intervention group patients. No gold standard exists for pain assessment in sedated and ventilated patients.
Time Frame: Within 24 hours of Enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 16 | 14
Participants | 0 | 0

17. Other Pre Specified Outcome: Expected Adverse Event Related to Device- Thrombophlebitis
Description: Thrombophlebitis assessed as symptomatic non central nervous system venous or arterial thrombus documented radiographically or ultrasonographically in the upper extremity to which the study intervention was applied.
Time Frame: Within 1 week of Enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 16 | 14
Participants | 0 | 0

18. Other Pre Specified Outcome: Expected Adverse Event Related to Device- Sepsis
Description: Sepsis assessed within one week of index arrest as either i) the presence of microbiologically proven, clinically proven, or suspected infection; or ii) presence of Systemic Inflammatory Response Syndrome (SIRS); and iii) development of at least one organ dysfunction within the preceding 24 hours.
Time Frame: Within 1 week of Enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 16 | 14
Participants | 0 | 0

19. Other Pre Specified Outcome: Expected Adverse Event Related to Cardiac Arrest
Description: Related to Cardiac Arrest The following are commonly observed in patients who experience cardiac arrest, and may or may not be attributable to specific resuscitation therapies. These will be monitored and reported but not classified as serious adverse events. Clinical diagnoses of pneumonia, cerebral bleeding, stroke, seizures, bleeding requiring transfusion or surgical intervention, rearrest, pulmonary edema, serious rib fractures, sternal fractures, internal thoracic or abdominal injuries as noted in the hospital discharge summary.
Time Frame: Discharge or 30 days after index arrest
Population: Participants were included in this analysis if they survived to discharge. Also excluded were 3 participant (all from the control group) with missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 7 | 3
Participants | 6 | 3

20. Other Pre Specified Outcome: Unexpected Adverse Event
Description: These will be defined as any serious unexpected adverse effect on health or safety or any unexpected life-threatening problem caused by, or associated with, a device, if that effect or problem was not previously identified in nature, severity, or degree of incidence in the investigation plan or application, or any other unexpected serious problem associated with a device that relates to the rights, safety or welfare of subjects. Death or neurological impairment will not be considered an adverse event in this study, as it is an expected part of the natural history of the illness for a large proportion of the population.
Time Frame: Discharge or 30 days after index arrest
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 16 | 14
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days after cardiac arrest.
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 9/16 | 8/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 1/16 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=16) | Control Group (N=14)
Temporary occlusion of IV in the Emergency Department (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — A single patient (6%) in the intervention group had transient occlusion of their upper extremity intravenous line, which immediately resolved on repositioning of the blood pressure cuff.

LIMITATIONS AND CAVEATS:
This was a single-center pilot study. The rate of incomplete application of the intervention may be higher in a multi-center study. It lacked power to detect significant differences in outcomes, and did not include immunologic markers or markers of cardiac or brain injury. It assessed feasibility of the intervention rather than to assess whether RIC achieved a significant difference in biomarkers or clinical outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-08-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT04265807/Prot_000.pdf